CLINICAL TRIAL: NCT05450926
Title: Appropriate Sonoanatomical Approach in Ultrasound-guided Selective Cervical Root Block
Brief Title: Selective Cervical Root Block for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: Selective cervical root block
Record Dates: First submitted 2022-02-17; First posted 2022-07-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Neck Pain
Keywords: Sonoanatomy; Cervical nerve root block; Neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy volunteers (No Intervention): Two Algology Specialists will record the localization and number of cervical spinal nerve, transverse process cornes and surrounding vascular structures at cervical C4-5-6-7 levels in healthy volunteers by Doppler USG.
- patients with cervical radicular pain (Active Comparator): Two Algology Specialists will apply cervical root block to patients with cervical radicular pain guided by Doppler USG, and pain scores of the patients will be evaluated with VAS (visual analog scale) before and after the procedure.
  Interventions: Procedure: Ultrasound-guided selective cervical nerve root block
- human cadavers (Other): Seven formalin-containing human cadavers will be examined by 3 anatomy doctors at Ankara University Faculty of Medicine, Department of Anatomy to determine the morphology of the spinal nerve, vertebral artery, assending and deep arteries in the cervical foraminal region, as well as the radicular arteries.
  Interventions: Procedure: Ultrasound-guided selective cervical nerve root block

INTERVENTIONS:
Procedure: Ultrasound-guided selective cervical nerve root block — The volunteer will be placed in the lateral decubitus position with the examined side up and the ultrasonographic examination will be started. Using a high frequency 6-18 MHz linear transducer, scanning in the cephalad and caudal direction until the cervical tubercles are identified in the short axis of the vertebra at the cricoid level, the localization and number of the target nerve root and vascular structures in the foraminal opening between the anterior and posterior tubercles of the transverse process from C4 to C8. will be defined as Unlike healthy volunteers, local anesthetic and steroid injections will be administered to the target nerve.
  Arms: human cadavers; patients with cervical radicular pain

SUMMARY:
Currently, selective cervical nerve root injections are recommended under the guidance of fluoroscopy, ultrasonography and computed tomography in patients with chronic cervical radicular pain who do not respond to conservative treatments and are not planned for surgery. Various serious complications, mainly vascular, have been reported in the literature. These complications include vertebral artery injury, spinal cord and brain stem infarction. The arteries of the cervical spinal cord are the vertebral, ascending, and deep cervical arteries arising from the aorta.The arteries arising from these main arteries and reaching the intervertebral foramen are called segmental arteries, the arteries reaching the epidural region from the intervertebral foramen and the radicular arteries, and the branches reaching the spinal cord are called the medullary artery. These small arteries supplying the spinal cord lie close to the spinal nerve in the foramen between the anterior and posterior trabercules. Vasospasm or embolism, which occurs as a result of direct needle trauma to these vascular structures around the target nerve or injection of particulate steroids, are the most common causes of complication development.

The aim of our study is to identify the vascular structures around the foramen in selective cervical root injection, which has proven effectiveness in cervical radicular pain, to determine the most reliable method for positioning the needle while reaching the target nerve under US guidance and to prevent possible complications.

DETAILED DESCRIPTION:
A total of 50 healthy volunteers and 10 patients with cervical radicular pain, between the ages of 18-70, height above 155 cm and body mass index 25 and below, in the Algology Clinic of the University of Health Sciences Dışkapı Yıldırım Beyazıt Training and Research Hospital will be included in the study. Those who have structural disorders in the neck region and who have undergone neck surgery will not be included in the study. 7 cadavers will be included in the study in Ankara University Faculty of Medicine, Department of Anatomy.

2 Algology specialists from Health Sciences University Dışkapı Yıldırım Beyazıt Training and Research Hospital Algology Clinic and 3 doctors from Ankara University Medical Faculty Anatomy Department will participate in the study. Two Algology Specialists will record the localization and number of cervical spinal nerve, transverse process cornes and surrounding vascular structures at cervical C4-5-6-7 levels in healthy volunteers by Doppler USG. Again, two Algology Specialists will apply cervical root block to patients with cervical radicular pain guided by Doppler USG, and pain scores of the patients will be evaluated with VAS (visual analog scale) before and after the procedure. Seven formalin-containing human cadavers will be examined by 3 anatomy doctors at Ankara University Faculty of Medicine, Department of Anatomy to determine the morphology of the spinal nerve, vertebral artery, assending and deep arteries in the cervical foraminal region, as well as the radicular arteries.

Demographic characteristics (age, gender, BMI, body height) of 50 volunteers and 10 patients with cervical radicular pain will be recorded. The pain intensity of 10 patients with cervical radicular pain will be determined and recorded with the VAS (visual analog scale) score before the procedure and at 1,2,3 and 4 weeks after the procedure, by calling the patients for control.

The cadavers will be dissected after being placed in the supine position and bilaterally from C4 to C7. Neurovascular complexes will be defined.

Efforts will be made to determine the most appropriate needle pathway to reach the target cervical nerve.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers patients with cervical radicular pain

Exclusion Criteria:

Patients who have structural disorders in the neck region and who have undergone neck surgery

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the vascular structures around the needle pathway while approaching the nerve to be applied cervical spinal nerve block with a needle. | 15 days
  Will evaluate the vascular structures around each C5, C6, and C7 nerve root , with Doppler ultrasound imaging. The pain scores of the patients will be evaluated with VAS (visual analog scale) by applying cervical root block under the guidance of Doppler USG to patients with cervical radicular pain.

SECONDARY OUTCOMES:
VAS (visual analog scale) | 15 days
  Pre- and post-procedure pain scores of the patients will be evaluated with VAS (visual analog scale) by applying cervical root block under the guidance of Doppler USG to patients with cervical radicular pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, Study Director — Diskapi Yildirim Beyazit Education and Research Hospital; Ayhan Cömert, Study Director — Ankara University Faculty of Medicine; Damla Yürük, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Dişkapi Reserch and Education Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No